CLINICAL TRIAL: NCT03104127
Title: Effect of a Community-based, Bionic Leg Rehabilitation Program on Biomechanical, Cardiovascular and Performance Outcomes in Patients With Chronic Stroke
Brief Title: Effect of Using a Lower Limb Robotic Device for Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Hobbs Rehabilitation (Other); AlterG (Unknown); University of Gloucestershire (Other); University of Chester (Other); University of Southampton (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RKE_2017_001
Record Dates: First submitted 2017-03-02; First posted 2017-04-07 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Gait, Hemiplegic; Quality of Life; Vascular Stiffness; Stroke
Keywords: Lower-limb robotic device; Gait; Balance; Pressure; Chronic stroke; Blood pressure; Blood velocity; Aerobic fitness; Strength
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Alter G Bionic Leg (Experimental): Participants randomised to a group including normal therapy (physiotherapy) and the use of a Alter G robotic bionic leg. All participants have previously completed normal NHS therapy.
  Interventions: Device: Alter G Bionic Leg; Other: Normal therapy (physiotherapy)
- Normal therapy (Active Comparator): Participants randomised to a group including normal therapy (physiotherapy) only. All participants have previously completed normal NHS therapy.
  Interventions: Other: Normal therapy (physiotherapy)
- Usual care (No Intervention): Have completed normal NHS therapy and no longer (> 6 months) receive active physiotherapy.

INTERVENTIONS:
Device: Alter G Bionic Leg — Participants are randomized to a 10 week, community-based bionic leg programme. Participants must use the leg for a minimum of 1 hour per day and continue to have active physical therapy sessions.
  Arms: Alter G Bionic Leg
Other: Normal therapy (physiotherapy) — Participants are randomized to a normal therapy (physiotherapy) only program. Participants are also advised to undertake 1 hour a day of physical activity and have active physical therapy (physiotherapy) sessions.
  Arms: Alter G Bionic Leg; Normal therapy

SUMMARY:
This study will investigate if a lower limb robotic device can be used in a community setting to increase the amount of physical activity that individuals undertake following stroke and consequently improve biomechanical, physiological and health outcomes, in patients with stroke.

DETAILED DESCRIPTION:
Recent advances in technology have helped to develop robotic devices to aid gait training in order to develop more normal movement patterns, strengthen the quadriceps and improve quality of gait. Lower limb robotic devices have been shown to increase functional mobility, walking speed, step length, balance and endurance within a clinical setting. The purpose of this study is to see if a lower limb robotic device leg can be used in a community setting to improve biomechanical (gait, balance, lower-limb strength), physiological (vascular health) and performance outcomes (aerobic fitness, strength) in patients with chronic stroke

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of stroke within 3-60 months
* Community patients that are medically stable and currently receiving therapeutic input from Hobbs Rehabilitation
* Individuals who are able to stand and step with an aid or assistance
* Cognitively aware of task demands
* Height: 5ft 2-6ft 3 (158-192 cm)
* Weight: <25 stone (< 159kg)

Exclusion Criteria:

* Unresolved deep vein thrombosis
* Unstable cardiovascular conditions
* Open wounds
* Active drug resistant infection
* Recent fractures of involved limb
* Peripheral arterial disease
* Incontinence
* Severe osteoporosis
* Non weight bearing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Gait analysis at 10-weeks post-intervention | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each gait analysis assessment will take 30 minutes
  Eight Qualisys cameras (six Oqus 3+, two Oqus 5+, Goteborg, Sweden) will be used to measure joint angles, rotations, hip obliquity, segment accelerations and velocities. Six Degrees or Fredom 6DoF 27 point marker set will be used and joint centres identified through palpation. The participants will be asked to walk for 6 meters for minimum of three trials in order to obtain walking gait patterns.
Change from baseline Gait analysis at 10-weeks post-intervention | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each gait analysis assessment will take 30 minutes
  The participants will be asked to walk for 6 meters, over a pressure mat (RSscan Footscan, Ipswitch, UK), for minimum of three trials in order to obtain walking gait patterns.
Change from baseline Gait analysis at 10-weeks post-intervention | aseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each gait analysis assessment will take 30 minutes
  A BTS G-Walk (Brooklyn, New York) sensor will also be worn by the participants to collect additional spatio-temporal gait parameters(cadence, speed, stride/step length, stance/swing phase duration, single/double support duration and pelvic girdle angles).

SECONDARY OUTCOMES:
Timed-up-and-go | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. The timed-up-and-go assessment will take 10 minutes
  A BTS G-walk system will be used to collect Timed-Up-and-Go data. From a seated position, participants will stand, walk to a cone 3 m away, walk around the cone, and walk back to the chair sit back down. Participants will complete two familiarisation trials prior to the actual test itself. A minimum of three trials will be performed
Ashworth scale | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 10 minutes
  An adapted Modified Ashworth Scale will be used to assess muscle function. This will include the assessment of; Hip flexion, extension, abduction, adduction; Knee flexion, extension; Ankle dorsiflexion, plantar flexion. Each movement will be graded from 0-5.
Body mass | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 5 minutes
  Body weight and body mass index will be measured
Central and peripheral blood pressures | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 5 minutes following 20 minutes supine rest.
  Pulse wave analysis (PWA) will investigate central blood pressures, augmentation index and arterial stiffness following 20 minutes supine rest. Pulse wave velocity (PWV) will also be recorded between the carotid (right and left) and femoral artery.
Arterial stiffness and blood velocity of the carotid artery | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 5 minutes following 20 minutes supine rest.
  Following 20 minutes supine rest, local arterial stiffness of the right and left carotid arteries will be imaged 1-2 cm proximal to the bifurcation using B-mode ultrasound.Doppler ultrasonography will be used to calculate bilaterally volumetric blood flow in the carotid artery. Blood flow will be recorded using a Doppler spectral trace for 1 minute during supine rest.
Physical fitness | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 6 minutes.
  A 6-minute shuttle walk test will determine total distance walked. Participants' perception of exertion will be measured at 2, 4 and 6 minutes.
Strength | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each assessment will take 15 minutes.
  Lower Limb muscle strength will be assessed using a Lafayette hand held dynamometer (Lafayette, USA). Measures will include; Hip abduction, adduction, flexion; Knee flexion, extension;. Ankle dorsiflexion, plantar flexion. Participants will be on a massage bed and perform up to three maximal trials for each measure with a minimum of one minutes rest between each measure.
7-day physical activity | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up.
  An ActivPal physical activity monitor will be used for 7 days at baseline, 5 weeks into the intervention, and on completion of the 10 week intervention to assess participants daily physical activity. Measures include; time seated, time standing, ambulation, number of steps, number of sit to stands, and energy expenditure.
Postural Sway | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up. Each postural sway analysis assessment will take 20 minutes
  Postural sway parameters will be calculated on the basis of centre of pressure. Time series will be acquired by means of a pressure mat mounted on top of a Kistler force platform (Kistler, Winterthur, Swizerland). Participants will stand on the pressure mat, unaided if possible, and trials will consist of eyes open shoes on, eyes closed shoes on, eyes open shoes off, eyes closed shoes off. A minimum of three trials will be performed for each condition, each lasting 10s
Manual Muscle Test | Baseline, 10-week post-intervention, 3 month follow-up, 12 month follow-up. Each assessment will take 5 minutes
  This will include the assessment of; Hip flexion, extension, abduction, adduction; Knee flexion, extension; Ankle dorsiflexion, plantar flexion on a 5-point scale. The function of the muscle will be graded from 0 (no contractions felt in the muscle) to 5 (holds test position against strong pressure).

OTHER OUTCOMES:
Dynamic gait index | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  8-item test that assesses dynamic balance and gait ability. Scored by rating the participants performance; walking on a level surface, changing speed while walking, turning the head from side to side and up and down while walking, sudden turns, obstacle negotiation, and stair negotiation. The dynamic gate index has excellent reliability (ICC > 0.94; Lin et al., 2010) and validity (r = 0.83; Jonsdottir & Cattaneo, 2007).
Berg Balance | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  14-item test that assesses static and dynamic balance ability and fall risk in adult populations. Each activity is scored from 0-4, determined by the ability to perform the assessed activity with an overall maximum score of 56. The Berg Balance scale has excellent reliability (ICC > 0.95) and strong correlations with the Fugl-Meyer and Postural Assessment Scale for Stroke patients (r > 0.90).
Balance Confidence Scale | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  16-item self-report measure in which patients rate their balance confidence when performing various ambulatory activities. Rated from 0-100. This scale has excellent test-retest reliability (ICC = 0.85) within the Stroke population and adequate correlations with the Functional Gait Assessment (r = 0.53) in community dwelling elderly (Winsley & Kumar, 2010).
Walking Ability Questionnaire | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  19-item questionnaire to assess the participant's social limitations resulting from decreased walking ability. Mobility is classified as independent, supervised, assisted, wheelchair or unable for 19 ambulatory activities commonly performed in the home (8) and community (11).
Functional Ambulation Classification | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  Assesses functional ambulation in participants undergoing physical therapy. Ranges from non-functional walking to independent walking outside with a scale for 0-5 respectively. The Functional Ambulation Classification has excellent validity with the 6 minute walking test in acute Stroke patients
International Physical Activity Questionnaire | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  Collects information on the time spent (number of days and average time per day) spent being physically active.
Older Peoples Quality of Life Questionnaire | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  36-item questionnaire that assesses quality of life. Each question is rated from 0-5 from very bad to very good respectively. Previously this has shown to have excellent test-retest reliability (ICC = 0.92) and has features that made it a more suitable outcome measure of QOL in older people compared with the frequently used measure, the SF-12. 36-item questionnaire that assesses quality of life. Each question is rated from 0-5 from very bad to very good respectively. Previously this has shown to have excellent test-retest reliability (ICC = 0.92) and has features that made it a more suitable outcome measure of QOL in older people compared with the frequently used measure, the SF-12. 36-item questionnaire that assesses quality of life. Each question is rated from 0-5 from very bad to very good respectively.
Trail Making | Baseline, 10-week post-intervention, 3-month follow-up, 12 month follow-up
  A neuropsychological test of visual attention and task switching. Consists of two tests, including: i) a test in which the participant is instructed to connect 25 numerical dots in order, and ii) a test in which the participant is instructed to connect 25 numerical and alphabetical dots in order.

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- University of Winchester, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faulkner J, Wright A, Stone K, Fryer S, Martinelli L, Lambrick D, Paine E, Stoner L. Effect of home-based, overground robotic-assisted gait training on vascular health in people with chronic stroke. Front Neurol. 2023 Mar 10;14:1093008. doi: 10.3389/fneur.2023.1093008. eCollection 2023. PMID 36970545